CLINICAL TRIAL: NCT02557529
Title: Progressive Resistance Training in Head and Neck Cancer Patients During Concomitant Chemoradiotherapy - The DAHANCA 31 Study
Brief Title: Progressive Resistance Training in Head and Neck Cancer Patients During Concomitant Chemoradiotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruition
Sponsor: Herlev Hospital (Other)
Collaborators: Aarhus University Hospital (Other); Odense University Hospital (Other); Danish Head and Neck Cancer Group (Network)
Responsible Party: Principal Investigator, Julie Gehl, M.D., Dr. Med. Sci., Herlev Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: DAHANCA 31
Record Dates: First submitted 2015-09-11; First posted 2015-09-23 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Head and Neck Neoplasms; Weight Loss
Keywords: Head and Neck Cancer; Concomitant chemoradiotherapy; Exercise Training; Progressive Resistance Training; Weight loss; Lean Body Mass; Body Composition
MeSH Terms: conditions — Head and Neck Neoplasms; Weight Loss | interventions — Exercise; Diet Records

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progressive Resistance Training (Experimental): 12 weeks progressive resistance training (PRT) during and after concomitant chemoradiotherapy. Also optional/voluntary physical activity performed on their own is registered, as well as diet diary.
  Interventions: Behavioral: Progressive Resistance Training; Behavioral: physical activity; Behavioral: Diet diary
- Control (Active Comparator): Control arm. Optional/voluntary physical activity performed on their own is registered, as well as diet diary.
  Interventions: Behavioral: physical activity; Behavioral: Diet diary

INTERVENTIONS:
Behavioral: Progressive Resistance Training — 12 weeks supervised resistance training program. Details of the program: 12 weeks, 3 sessions per week, 7 exercises in training machines (leg press, leg curl, hamstring curl, chest press, lateral pull down, sit-ups and back extensions). In general 2-3 sets of 8-15 repetitions will be performed following a progression plan starting with more repetitions at lower intensity progressing to fewer repetitions at higher intensity during the 12-week period (American College of Sports Medicine Position Stand)
  Arms: Progressive Resistance Training
Behavioral: physical activity — Weekly diary of performed physical activity using the Physical Activity Score (PAS) during the 12-weeks intervention
  Other Names: Diary of performed physical activity
Behavioral: Diet diary — Weekly diet diary during the 12-weeks intervention

SUMMARY:
72 patients with head and neck cancer, undergoing primary treatment with radiation therapy and concomitant weekly cisplatin, will be recruited to this multicentre trial.

Randomized 1:1 to either 12-week progressive resistance training (PRT) program or control arm, starting together with concomitant chemoradiotherapy (CCRT) Stratified by centre, gender, p16-status and body mass index (BMI) below or above 30.

Primary endpoint is difference in change in lean body mass (LBM) between the groups and the endpoint is reduction of LBM loss in intervention arm by 25% compared to control.

Secondary endpoints include side-effects to treatment, change in body composition, physical function and strength, and compliance to PRT. Questionnaires on QoL, diet, voluntary exercise and work affiliation will also be registered.

Blood samples for explorative analyses will be drawn and optional muscle biopsies drawn for proteomics analyses and histological analyses.

DETAILED DESCRIPTION:
The PRT program will start about the onset of radiotherapy. The program consists of 7 exercises in training machines and involves the major muscle groups of the body.

The program has previously been found to successfully restore the loss of lean body mass (LBM) in head and neck cancer patients post-treatment. A group based approach will be used to facilitate a social and motivating training environment for the patients. A pilot study (NCT02068950) showed feasibility of PRT during CCRT.

In addition to baseline data (height, tumor stage, performance status, etc), the following parameters will be registered: Weight, patient reported side effects, as well as a questionnaire on amount of physical activity and food intake.

Physical function and strength will be tested at baseline, after the course of chemoradiotherapy and at the end of the 12-week PRT programme, and at 6 and 12 months follow-up. DXA scans for body composition will be performed using a Lunar iDXA (GE Healthcare).

Blood samples will be drawn at regular intervals during the 12 weeks and at follow-up.

Patient reported quality of life (EORTC Quality of Life Questionnaire (QLQ)-C30 and QLQ-H&N35) will also be registered.

Muscle biopsies will be taken three times: at baseline, after treatment and after 12-weeks PRT.

Study duration is expected to be 18 months and an additional 12 months for follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy verified head and neck squamous cell carcinoma referred for primary curatively intended treatment.
* Candidates for concomitant chemoradiotherapy (2Gyx33-34; 6F/W; weekly cisplatin 40mg/m2, max. 70 mg/weekly) according to Danish Head and Neck Cancer Group (DAHANCA) guidelines (T1-4, N1-3, M0)

  * Performance status 0-1
  * At least 18 years of age.

Exclusion Criteria:

* BMI below 20.5
* diabetes
* corticosteroid treatment for other diseases
* Tonsillectomy within the last week before inclusion.
* hemoglobin below 6 mmol/l
* leucocytes below 2.5 x 10^9 /l
* thrombocytes below 50 x 10^9 /l
* comorbidities, social, familial or geographical conditions, that could compromise attendance or results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-08; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Change in LBM (lean body mass) | at 12-weeks post PRT
  change in kilograms

SECONDARY OUTCOMES:
Change in LBM (lean body mass) | at 6 weeks, and 6 and 12 months post RT
  change in kilograms
Fat mass | at 6 and 12 weeks, and 6 and 12 months post RT
  change in kilograms
Weight loss | at 6 and 12 weeks, and 6 and 12 months post RT
  in kilograms
Patient reported pain | at 6 and 12 weeks, and 6 and 12 months post RT
  Measured by NRS-scale
Patient reported Quality of Life | at 6 and 12 weeks, and 6 and 12 months post RT
  QLQ-C30 questionnaire
Muscle strength | at 6 and 12 weeks, and 6 and 12 months post RT
  measured using chest press and leg press
Chair rise | at 6 and 12 weeks, and 6 and 12 months post RT
  measured using 30 s. chair rise
arm curls | at 6 and 12 weeks, and 6 and 12 months post RT
  measured using 30 s. arm curls
Stair climb | at 6 and 12 weeks, 6 and 12 months
  steps/sec
Compliance to PRT program | at 12 weeks post PRT
  No. of attended sessions out of total
Physical activity | at 6 and 12 weeks, and 6 and 12 months post RT
  measured by PAS (physical activity scale)
Percent of patients with feeding tubes | at 6 and 12 weeks, and 6 and 12 months post RT
Resumption of work | At 12 months follow-up
  No. of days from end of radiotherapy until back at work at full time (or the hours of work per week as before therapy)
Percent relapses | at 12 months follow-up
  Percent of patients having relapse within 12 months after radiotherapy
Cytokines | at 3, 6, 8, 10, and 12 weeks
  Measurement of different cytokines, changes over time and after bout of PRT. Will be measured regularly during the 12 weeks of PRT.
Muscle biopsies | at 6 and 12 weeks, and at 12 months follow-up
  protein will be measured using the proteomic approach. Muscle fiber type and size will be evaluated.
Patient satisfaction | at 12 weeks
  Study specific questionnaire regarding pros and cons of attending the study
NK-cells | at 3 and 12 weeks
  Measuring NK-cells. NK-cells may increase after exercise and show tumor inhibiting effect.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Gehl, Principal Investigator — Herlev Hospital
Locations (1):
- Department of Oncology, Copenhagen University hospital, Herlev, Herlev, Denmark

REFERENCES:
- [Background] Lonkvist CK, Lonbro S, Vinther A, Zerahn B, Rosenbom E, Primdahl H, Hojman P, Gehl J. Progressive resistance training in head and neck cancer patients during concomitant chemoradiotherapy -- design of the DAHANCA 31 randomized trial. BMC Cancer. 2017 Jun 3;17(1):400. doi: 10.1186/s12885-017-3388-0. PMID 28578654